CLINICAL TRIAL: NCT01366352
Title: Pharmacokinetics and Bioavailability Comparison of Two Different Formulations of MNTX Tablets: A Double-Blind, Single Dose, Crossover, Phase 1 Study in Normal Volunteers
Brief Title: Pharmacokinetics and Bioavailability Comparison of Two Different Formulations of MNTX Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNTX 1202
Record Dates: First submitted 2011-05-27; First posted 2011-06-06 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Normal Volunteers
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): MNTX tablet
  Interventions: Drug: MNTX tablet (Formulation 1)
- Arm 2 (Experimental): MNTX tablet
  Interventions: Drug: MNTX tablet (Formulation 2)

INTERVENTIONS:
Drug: MNTX tablet (Formulation 1)
  Arms: Arm 1
Drug: MNTX tablet (Formulation 2)
  Arms: Arm 2

SUMMARY:
This was a single-center, double-blind, randomized, cross-over Phase 1 study in normal, healthy volunteers. Study treatment entailed single doses of two different formulations of MNTX tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Weight between 55 and 85 kg
2. In good health, based on history, physical examination, and appropriate laboratory and diagnostic tests at screening, with no evidence of clinically significant chronic medical condition
3. Non-smokers.

Exclusion Criteria:

1. History of evidence of cardiovascular, gastrointestinal, hepatic, musculoskeletal, neurological, pulmonary, renal, or other significant chronic illness
2. History of asthma, allergic skin rash, significant allergy, or other immunologic disorder
3. Consumption of barbiturates or other inducers or inhibitors of CYP450
4. History or suspicion of alcohol or drug abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-02; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of MNTX administered as two different oral formulations | 7 days
  To determine and compare the plasma pharmacokinetics and extent of single, oral doses of two different oral formulations of MNTX in normal healthy volunteers.

SECONDARY OUTCOMES:
Half-life of MNTX administered as two different oral formulations | 7 days
  To determine and compare the plasma pharmacokinetics and extent of single, oral doses of two different oral formulations of MNTX in normal healthy volunteers.
Time from a single dose to maximum concentration (Tmax) of MNTX administered as two different oral formulations | 7 days
  To determine and compare the plasma pharmacokinetics and extent of single, oral doses of two different oral formulations of MNTX in normal healthy volunteers.
Area under the plasma concentration (AUC) of MNTX administered as two different oral formulations | 7 days
  To determine and compare the plasma pharmacokinetics and extent of single, oral doses of two different oral formulations of MNTX in normal healthy volunteers.
Total body clearance over bioavailability (CL/F) of MNTX administered as two different oral formulations | 7 days
  To determine and compare relative bioavailability, and extent of single, oral doses of two different oral formulations of MNTX in normal healthy volunteers.
Volume of distribution over bioavailability (V/F) of MNTX administered as two different oral formulations | 7 days
  To determine and compare the plasma pharmacokinetics, relative bioavailability, and extent of single, oral doses of two different oral formulations of MNTX in normal healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States